CLINICAL TRIAL: NCT03454178
Title: Sensitivity, Specificity, and Positive and Negative Predictive Values of Automatic Office Blood Pressure Measurement and Traditional Office Blood Pressure Measurement in a Chinese Population
Brief Title: Accuracy of AOBP in a Chinese Population
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lee Kam Pui, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: CUHK-188
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2020-09

CONDITIONS: Hypertension
Keywords: AOBP; ABPM
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hypertensive patients: 150 Chinese patients with a diagnosis of essential hypertension from a primary care clinic
  Interventions: Diagnostic Test: WatchBP Office (BP measurement machine)

INTERVENTIONS:
Diagnostic Test: WatchBP Office (BP measurement machine) — BP measurement: The nurse or assistant will leave the room after confirmed validity and the WatchBP will automatically measure BP for the participant at 1-minute intervals for 3 more readings; previous research showed that accurate BP readings could be obtained using 1-minute intervals. This is also the measuring method suggested by the manufacturer. The machine will automatically calculate the mean BP using the 3 readings. The mean BP value will be used for analysis. The diagnostic cutoff for diagnosing HT will be ≥135/85 for AOBP

SUMMARY:
Background: Traditional office blood pressure (BP) measurement is often inaccurate and is inferior to out-of-office measurements, such as ambulatory blood pressure monitoring (ABPM), in predicting cardiovascular outcomes. A relatively new BP measurement method, called Automatic Office Blood Pressure measurement (AOBP), may provide similar BP readings to ABPM (latest clinical gold standard for BP measurements) and can easily be conducted in clinics. AOBP machines measure BP repeatedly 3-5 times with 1-min intervals and automatically provide the mean BP value. While AOBP was used in landmark trials (e.g. SPRINT trial) and was shown to eliminate white-coat effect, AOBP is rarely used in Hong Kong partly because there is no data concerning the accuracy of AOBP in Chinese. Almost all previous AOBP research used BpTRU (AOBP model), but BpTRU manufacturer was shut down permanently.

Aim: To assess if WatchBP Office (another AOBP model) has superior diagnostic accuracy than traditional office BP measurements, when compared to ABPM readings.

Method: 150 Chinese adult patients with a diagnosis of essential hypertension will be recruited consecutively from a Government-funded primary care clinic. All patients will have their BP measured by a 48-hour ABPM, a WatchBP office, and two traditional office blood pressure measurements.

ABPM will be considered the gold standard; sensitivity, specificity, positive and negative predictive values of AOBP and traditional BP to diagnose elevated BP level, masked hypertension and white-coat hypertension will be calculated and compared

Implication: if WatchBP provides closer BP readings to ABPM, this can lead to its implementation in routine clinical practice

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of essential hypertension

Exclusion Criteria:

* (i) severe hypertension as defined by clinical systolic BP ≥180 mmHg and/or diastolic BP ≥110 mmHg (because they may need emergency treatment and it is unethical to delay such treatment due to the proposed project), (ii) inability to provide consent, (iii) pregnancy, (iv) night-time occupations (we need to compare AOBP and clinic BP readings to daytime ABPM average when the patient should be awake), (v) are occupational drivers (because potential dangers in driving could occur when patients are asked to remain still), (vi) receiving anti-coagulants (to prevent bruises when using ABPM), (vii) with known atrial fibrillation (as ABPMs and AOBP use have not been validated in this group)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertensive patients in primary care
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2019-12-29 (Actual); Study Completion 2019-12-29 (Actual)

PRIMARY OUTCOMES:
compare BP readings from AOBPs, ABPM, and traditional office BP | 1 year
  mean difference of systolic BP (SBP) and diastolic BP (DBP) between AOBP machines (WatchBP Office, BpTRU)/office BP and daytime ABPM will be compared by the two-tailed t-test; A Bland-Altman type plot will be shown for both comparisons. Pearson correlations will be used to compare mean readings of office BP, AOBP and daytime ABPM.

SECONDARY OUTCOMES:
sensitivity/specificity, positive and negative predictive value of AOBP vs traditional BP measurement | 1 year
  sensitivity/specificity, positive and negative predictive value of diagnosing elevated BP, masked hypertension, and white-coat hypertension of AOBP and office BP will be compared using ABPM as the gold standard

CONTACTS AND LOCATIONS:
Locations (1):
- Lek Yuen Clinic, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Will be willing to share on request